CLINICAL TRIAL: NCT01326897
Title: Healthy Homes/Healthy Families
Acronym: HHHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Cancer Coalition of South Georgia (Unknown)
Responsible Party: Principal Investigator, Michelle C. Kegler, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00048222; HHHF (Other: Other)
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Diseases
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison Group (Active Comparator): Comparison group participants will be given health education materials.
  Interventions: Behavioral: Health Education
- Intervention' (Experimental): This group will receive the intervention (Healthy Homes/Healthy Families) as described below.
  Interventions: Behavioral: Healthy Homes/Healthy Families

INTERVENTIONS:
Behavioral: Healthy Homes/Healthy Families — Participants in the intervention group will work with coaches to make their homes more supportive of healthy eating and physical activity. Each intervention participant will receive a tailored home environment profile, and will select from a "menu" of healthy actions to make changes in their home. The intervention will be delivered over the course of 5 months, with 3 home visits, 4 coaching calls, and 4 support mailings.
  Arms: Intervention'
Behavioral: Health Education — Study participants in this group will receive health education materials by mail (3 times over the course of 5 months).
  Arms: Comparison Group

SUMMARY:
The purpose of the study is to learn how to make homes more supportive of healthy eating and physical activity. As part of the study, participants will be randomly assigned to one of two groups. One group will receive materials with information on healthy eating and physical activity. The materials will be mailed 3 times over a 5 month period. The other group will work with a coach to make their homes more supportive of healthy eating and physical activity. Working with a coach involves 3 home visits and 4 coaching telephone calls over a 5 month period. This group will also receive materials by mail 4 different times. All participants will be asked to complete 7 telephone interviews over a 1 year period. Participants will also be asked to wear an accelerometer, a small portable device that tracks movement from physical activity, for 7 days at 2 different points in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 35-65 years old
* BMI greater than or equal to 25
* Speak English
* Must live with at least one other person
* Live within 30 miles of 1 of 9 clinics referring patients in the study
* Must have no contraindications for physical activity
* Must have no contraindications for participating in a medically unsupervised study

Exclusion Criteria:

* 1 person per household

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Diet & Physical Activity | Baseline, 6 months, and 12 months
  Diet and physical activity will be assessed by telephone interviews. Physical activity will also be assessed using accelerometers at baseline and 6 months.

SECONDARY OUTCOMES:
Weight | Baseline, 6 months, and 12 months
  Self-report weight will be assessed by telephone interview.
Changes in the home physical and social environment | Baseline, 6 months, and 12 months
  A home environment survey will be administered by telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Kegler, DrPH, MPH, Principal Investigator — Emory University, Rollins School of Public Health; Julie Gazmararian, PhD, Principal Investigator — Emory University, Rollins School of Public Health

REFERENCES:
- [Result] Kegler MC, Haardorfer R, Alcantara IC, Gazmararian JA, Veluswamy JK, Hodge TL, Addison AR, Hotz JA. Impact of Improving Home Environments on Energy Intake and Physical Activity: A Randomized Controlled Trial. Am J Public Health. 2016 Jan;106(1):143-52. doi: 10.2105/AJPH.2015.302942. PMID 26696290
- [Derived] Haardorfer R, Alcantara IC, Patil D, Hotz J, Kegler MC. Physical activity profiles of overweight and obese women in rural Georgia. JAMA Intern Med. 2014 Jan;174(1):148-9. doi: 10.1001/jamainternmed.2013.11571. No abstract available. PMID 24145657